CLINICAL TRIAL: NCT04550871
Title: A Pilot Study Investigating the Detection of Episodes of Significant Patient-Ventilator Asynchrony in Mechanically Ventilated Patients
Brief Title: A Pilot Study Investigating the Detection of Episodes of Severe Patient-Ventilator Asynchrony
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Autonomous Healthcare, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: S-101
Record Dates: First submitted 2020-09-03; First posted 2020-09-16 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Respiratory Failure
Keywords: Patient-ventilator asynchrony
MeSH Terms: conditions — Respiratory Insufficiency; Patient-Ventilator Asynchrony

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The goal of this study is to determine what percent of severe patient-ventilator asynchrony is detected in mechanically ventilated patients in the adult ICU and to determine delays in detecting those asynchronies by the staff that were correctly identified, and whether asynchrony status recorded during intermittent assessments by respiratory therapists is representative of periods in between such assessments.

DETAILED DESCRIPTION:
This is a prospective observational study. All decisions about ventilator settings, mode of ventilation, and sedative doses are determined by the critical care team attending to the patient. Patients will be enrolled within 6 hours after intubation and will be studied continuously until extubation. Patients will be monitored for asynchrony using Syncron-E tablets provided by Autonomous Healthcare. However, clinical staff will be blinded to the results of the tablet, and hence, there will be no change to clinical care.

Asynchrony index (which captures the fraction of breaths with asynchrony) will be calculated every minute by the Syncron-E tablet. The assessment of respiratory therapists at the time of ventilator checks will also be recorded including the following information: i) entering/exiting the room , ii) existence of a severe asynchrony episode based on the respiratory therapist's assessment and its type. Clinical staff will record the start of any severe asynchrony episode that they detect. Data related to the administrations of sedatives and anesthetics as well as major interventions (excluding any PHI) will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring intensive care unit admission
* Patients requiring invasive mechanical ventilation expected to last more than 24 hours
* Patients ventilated on PCV, PSV, VCV, or VC+ ventilation modes

Exclusion Criteria:

* Any patient not meeting inclusion criteria.
* Any patient receiving muscle relaxant (paralytics) for more than 24 hours.
* Any patient receiving inverse ratio ventilation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated in the intensive care unit
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of asynchrony events per minute and the asynchrony index | Up to 4 weeks
  The endpoints will be calculated starting from the end of each ventilator check (when the respiratory therapist is leaving the room) and cover the time from that time point until 5-minutes prior to the next ventilator check event. The endpoints will also be separately calculated for the 5-minute period immediately preceding the next ventilator check.

SECONDARY OUTCOMES:
Time difference between when the Syncron-E tablet detects the start of severe asynchrony episodes and when the clinician-detects the start of severe asynchrony episodes | Up to 4 weeks
Number of Syncron-E tablet-detected severe asynchrony episodes that went undetected by clinicians and the number of clinician-detected severe asynchrony episodes undetected by Syncron-E tablet | Up to 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Northeast Georgia Medical Center, Gainesville, Georgia, United States